CLINICAL TRIAL: NCT07296562
Title: Expert Consensus on the Use of Nutraceuticals in Pregnancy: A Delphi Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Nutriceuticals in Pregnancy
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Nutraceuticals; Pregnancy
Keywords: nutraceuticals; Pregnancy; Maternal Health; Fetal Health; Consensus; Delphi

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: The study population will consist of a purposive sample of experts in obstetrics, maternal-fetal medicine, and clinical nutrition who are actively involved in the care of pregnant patients and have experience or knowledge regarding the use of nutriceuticals in pregnancy.

SUMMARY:
This study is a Delphi-based expert consensus project aimed at developing evidence-informed recommendations for the safe and effective use of nutriceuticals during pregnancy. Despite widespread use of vitamins, minerals, and other dietary supplements in prenatal care, significant variability exists in clinical practice regarding indications, dosing, timing, and safety monitoring.

DETAILED DESCRIPTION:
This study is a non-interventional, methodological Delphi consensus project designed to develop standardized recommendations for the use of nutriceuticals during pregnancy. Nutriceuticals, including vitamins, minerals, antioxidants, omega-3 fatty acids, and herbal supplements, are commonly used to support maternal health and fetal development. However, evidence regarding optimal dosing, timing, and safety profiles is inconsistent, and practice patterns vary globally.

A steering committee of experts in obstetrics, maternal-fetal medicine, and clinical nutrition will conduct a thorough literature review and draft initial statements addressing key domains:

Indications for nutriceutical use (routine supplementation, deficiency prevention, high-risk pregnancies)

Recommended dosing and timing for common nutriceuticals (folic acid, iron, vitamin D, iodine, omega-3 fatty acids, etc.)

Safety considerations and contraindications (including herbal and non-standard supplements)

Monitoring strategies for maternal and fetal safety

Integration with dietary and lifestyle interventions

Counseling and patient education

A panel of experts in obstetrics and maternal nutrition will participate in multiple Delphi rounds. Panelists will rate each statement on a Likert scale for agreement. After each round, anonymized feedback will be provided, and statements not reaching the predefined consensus threshold (e.g., ≥70-80%) will be revised for subsequent evaluation.

The final output will consist of consensus-based recommendations for nutriceutical use in pregnancy, highlighting areas of strong agreement, areas of uncertainty, and research priorities. These recommendations aim to support safe, evidence-informed clinical practice for maternal and fetal health.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified obstetricians, maternal-fetal medicine specialists, or clinical nutritionists with ≥5 years of relevant clinical experience.

Active involvement in prenatal care and experience or knowledge in nutriceutical use during pregnancy.

Engagement in clinical teaching, research, guideline development, or professional society activities related to maternal health or nutrition.

Willingness and availability to participate in all Delphi rounds.

Provision of informed consent to participate.

Exclusion Criteria:

* Non-obstetric or non-nutrition specialty.

Less than 5 years of relevant clinical experience.

Limited or no experience with nutriceutical counseling/prescribing in pregnancy.

Significant undisclosed conflict of interest related to nutriceutical products.

Inability or unwillingness to participate in all Delphi rounds.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: he study population will consist of a purposive sample of experts in obstetrics, maternal-fetal medicine, and clinical nutrition who are actively involved in prenatal care and have experience or knowledge regarding the use of nutriceuticals in pregnancy.
  Panel Size and Rationale:
  Target enrollment: 20-35 experts.
  Sufficient to capture diverse perspectives while remaining feasible for multiple Delphi rounds.
  Minimum for analysis: 15 panelists, ensuring representativeness in case of attrition.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 6-12 weeks
  Level of expert consensus on statements regarding nutraceutical use in pregnancy, measured as the proportion of panelists reaching the predefined agreement threshold (e.g., ≥70-80%) for each statement across Delphi rounds.

SECONDARY OUTCOMES:
Secondary outcome | 6-12 weeks
  Consensus on indications for specific nutriceuticals (e.g., folic acid, iron, vitamin D, omega-3 fatty acids, iodine, herbal supplements).
  Consensus on optimal dosing, timing, and duration of supplementation.
  Consensus on safety monitoring protocols, including laboratory assessments and maternal/fetal surveillance.
  Consensus on contraindications and risk mitigation strategies for nutriceutical use.
  Consensus on integration with dietary and lifestyle interventions.
  Identification of areas of uncertainty requiring further research.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged